CLINICAL TRIAL: NCT00002936
Title: Hexamethylamine and VP-16 an Oral Regimin for HIV Malignancies: A Phase I/II Trial
Brief Title: Altretamine and Etoposide in Treating Patients With HIV-Related Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: DS 95-05; RPCI-DS-95-05; NCI-G97-1165
Record Dates: First submitted 1999-11-01; First posted 2004-05-13 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-02

CONDITIONS: Lymphoma; Sarcoma
Keywords: AIDS-related Kaposi sarcoma; recurrent Kaposi sarcoma; AIDS-related peripheral/systemic lymphoma
MeSH Terms: conditions — Lymphoma; Sarcoma; AIDS-related Kaposi sarcoma; Sarcoma, Kaposi | interventions — Altretamine; Etoposide

INTERVENTIONS:
Drug: altretamine
Drug: etoposide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of altretamine plus etoposide in treating patients with HIV-related cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine toxic effects of repeated courses of altretamine plus etoposide at the maximum tolerated dose (MTD). II. Assess the response duration and time to progression at the MTD in the treatment of HIV malignancies. III. Assess the efficacy of the combination on the immune systems of these individuals. IV. Assess the effect of the combination on the quality of life in these individuals.

OUTLINE: Patients are treated with altretamine (HMM) and etoposide for 2 weeks followed by 2 weeks of rest. This cycle is repeated for a minimum of 2 and a maximum of 6 cycles if there is no progression of disease. Patients who are in complete remission receive an additional 2 cycles (total of 8 cycles). There are different cohorts consisting of 4 patients each in which toxic effects will be evaluated with escalating doses of this combination. The MTD is defined as the dose level immediately below that at which half of the patients experience dose-limiting toxicity. Patients are followed for relapse and survival.

PROJECTED ACCRUAL: 20 patients will be accrued in 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Documented HIV antibody positive Histologically confirmed, by biopsy, non-Hodgkin's lymphoma that is in complete remission or stable/partial remission for a minimal period of one month And/or Histologically confirmed, by biopsy, Kaposi's sarcoma without stable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Hematopoietic: Absolute neutrophil count at least 500/mm3 Platelet count greater than 25,000/mm3 (unless secondary to lymphoma) Hepatic: Transaminases less than 5 times upper limit of normal AND Bilirubin less than 2.0, unless secondary to lymphoma Renal: Creatinine less than 2.0 mg/dL OR Creatinine clearance at least 60 mL/min Dose reduction of 21% if creatinine clearance 10-50 mL/min Dose reduction of 50% if creatinine clearance less than 10 mL/min Cardiovascular: No active cardiac arrhythmia or angina Pulmonary: Must exclude Pneumocystis carinii pneumonia if there is any suspicion of infection Other: No uncontrolled infections Not pregnant or nursing Adequate contraception for fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Patients with concurrent antiretroviral therapy should be on a stable dose of that therapy for at least one month prior to entry No concurrent cytotoxic chemotherapy Endocrine therapy: No concurrent hormone therapy Radiotherapy: No concurrent radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-07; Primary Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence P. Leichman, MD, Study Chair — Albany Medical College
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States